CLINICAL TRIAL: NCT03629379
Title: Response to Ustekinumab for Anti-tnf Induced Psoriasiform Skin Lesions
Acronym: STRAUSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S61472
Record Dates: First submitted 2018-05-14; First posted 2018-08-14 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2018-04

CONDITIONS: Inflammatory Bowel Diseases; Psoriasis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Psoriasis | interventions — Ustekinumab; Blood Specimen Collection; vedolizumab

STUDY DESIGN:
Intervention Model Description: prospective, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ustekinumab arm (Active Comparator): First 10 patients who are switched from anti-TNF to ustekinumab because of psoriasiform skin lesions refractory to 12 weeks of topical therapy.
  Interventions: Drug: Ustekinumab
- vedolizumab arm (Active Comparator): First 10 patients who are switched from anti-TNF to vedolizumab because of psoriasiform skin lesions refractory to 12 weeks of topical therapy.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Ustekinumab — Patients will receive standard dosing of ustekinumab with a single intravenous infusion of about 6mg/kg ustekinumab at week 0, followed by ustekinumab 90mg subcutaneously every 8 weeks.
  Other Names: Clinical disease activity of inflammatory bowel disease; Digital pictures of skin lesions; Scoring of (severity) of anti-TNF induced skin lesions; Skin biopsies; Blood sampling; Stool sampling
  Arms: ustekinumab arm
Drug: Vedolizumab — Patients will receive standard dosing of vedolizumab 300mg at weeks 0, 2, 6, and 14. Patients with Crohn's disease could receive an extra infusion at week 10.
  Other Names: Clinical disease activity of inflammatory bowel disease; Digital pictures of skin lesions; Scoring of (severity) of anti-TNF induced skin lesions; Skin biopsies; Blood sampling; Stool sampling
  Arms: vedolizumab arm

SUMMARY:
Using transcriptomics and proteomics to gain insights in the development of psoriasiform skin lesions under anti-tumor necrosis factor (TNF) therapy, and predicting response to ustekinumab.

DETAILED DESCRIPTION:
The investigators will prospectively include patients with Crohn's disease (CD) or ulcerative colitis (UC), who develop psoriasiform skin lesions (including psoriasiform eczema, psoriasis guttata, psoriasis inversa and pustulosis) under therapy with anti-TNF and refractory to at least 12 weeks of topical therapy. Since no scoring systems are available to describe (the severity of) anti-TNF induced skin lesions, the lesions will be followed up at different time points using 3 different methods. First, the Dermatology Life Quality Index (DLQI), which is a standardised questionnaire that is used in routine clinical practice to assess the impact of any type of skin lesion on the quality of life of the patient. Next a global visual analogue scale (VAS) to be filled out by the expert dermatologist based on the general appearance of the skin lesions, and finally a self-designed physician global assessment (PGA). Physician global assessment of paradoxical skin lesions will be based on the following:

* Number of body regions that are affected: 1 region (1 point), 2 or 3 regions (2 points) and more than 3 regions (3 points). The 8 regions to consider are: scalp, face, both axilla, groins, genital (including pubis and perineal), trunk (front and back + neck and collar), arms (including hands), legs (including feet)
* Location of skin lesions: face (1 point), palmoplantar (1 point), genital (1 point), flexural (1 point)
* Affected body surface area >10% (3 points)
* Presence of itching (1 point)
* Painful skin lesion (1 point)
* Is the lesion wet including erosions, pustules and maceration (2 points) or dry (0 points)?
* Is the lesion superinfected? Yes (1 point) or No (0 points)

The investigators plan to include 20 patients, namely the first 10 patients who will be switched to ustekinumab (UST, n=10, only available for patients with CD) and the first 10 patients who will be switched to anti-integrin therapy (VDZ, n=10). The latter will be used as a control group to evaluate whether starting ustekinumab or discontinuing anti-TNF leads to improvement of the lesions. Patients will be included through our outpatient clinic or infusion unit. The decision to start ustekinumab or vedolizumab will be based on routine clinical practice, and not be influenced by this study.

At the first evaluation (moment of treatment change), a blood draw (EDTA, serum, PAX gene) will be performed, the clinical CD or UC activity will be calculated by using patient reported outcome (PRO2) and Crohn's Disease Activity Index (CDAI) or Mayo score, and the patient will be asked to fill out a DLQI. Next, the patient will be send to one of two board certified dermatologists. The latter will document the skin lesions, take pictures of all lesions, state the clinical diagnosis and perform two punch biopsies of the affected skin ánd of unaffected skin at the contralateral sight. The dermatologist will also fill out the above mentioned VAS and PGA.

Patients switched to ustekinumab will receive standard induction with intravenous ustekinumab 6mg/kg, followed by subcutaneous ustekinumab 90mg every 8 weeks. Patients switched to vedolizumab will receive standard induction with intravenous vedolizumab 300mg at weeks 0, 2, 6, 10, 14 and every 8 weeks thereafter.

The patients will be re-evaluated 6-8 and 14-16 weeks after change in treatment. At week 6-8, patients will be clinically (including PRO2, CDAI/Mayo, and DLQI) and serologically (blood samples) re-evaluated by one of our three inflammatory bowel disease (IBD) specialists and all lesions will be photographed again. At week 14-16, re-evaluation by a gastroenterologist as well as dermatologist will take place. This will also include a new skin biopsy, but only at the initial site of the skin lesions (not the unaffected contralateral sight) (cfr. Study diagram). Dermatological response will be defined as a drop in VAS with at least 50%.

All blood samples will be analysed at the Translational Research in GastroIntestinal Disorders (TARGID) lab, Catholic University Leuven. One of the baseline skin biopsies will be send for histological examination by a certified pathologist (prof. dr. van den Oord) to obtain a correct histological diagnosis of the lesion. All the other biopsies will be stored in the TARGID-lab, Catholic University Leuven and will be used to perform transcriptomic and proteomic analyses (see further).

First, all patients included will be genetically characterize by using the Infinium Global Screening Array (GSA, Illumina). For the analyses the investigators will collaborate with the Department of Complex Genetics and Genomics Core Leuven. Next, a weighted polygenetic risk score will be calculated for all individuals. By performing a weighted risk score, the effect size and population frequency of the included genetic variants will be taken into account. The latter will be taken from already published genome-wide association studies. Using GSA will also enable the investigators to find new allele. Third, compare protein expression between the different patients groups will be compared by using serum tubes. Protein biomarkers in serum will be compared using the immunology panel (OLINK Proteomics). This panel is a high-throughput, multiplex immunoassay enabling analysis of 92 protein biomarkers across 96 samples simultaneously. The proteins will be analyzed following quality control and excluding markers with >75% missing data. To validate the found biomarkers the Mesoscale platform (Meso Scale Diagnostics) will be used. In addition, differences in gene expression in blood as well as skin biopsies will be compared. For the blood analyses PAX tubes will be used from the investigators' biobank. To extract RNA from PAX tubes the PAXgene Blood RNA Kit (Qiagen) will be used. For RNA extraction from skin biopsies AllPrep DNA/RNA Mini Kit (Qiagen) will be used. After extraction of RNA, next-generation single-end sequencing will be performed in collaboration with the Genomics core facility, Leuven. The high sequencing (4000NGS) platform from Ilumina will be used. Based on this proof of concept study a more limited panel of markers will be developed and evaluate in a confirmation cohort.

It is known that TNF, type I interferon (IFN) and interleukin-17 (IL-17) play an important role in the development of paradoxical psoriasiform skin lesions with the overproduction of IFN being the major driving force.(14, 33) However, the interplay between IL-17 and IFN is not clear. In addition, which immune cells are activated by IFN and through which cytokines is still unknown. To help solve these questions, skin biopsies will be used to further explore the interplay between IFN and other cytokines (IL-17, IL-22 and IL-23) and cells (innate lymphoid cells, ILC3) in patients treated with anti-TNF and how this interplay changes when treatment is changed to anti-IL12/23 therapy or vedolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD or UC, who develop psoriasiform skin lesions (including psoriasiform eczema, psoriasis guttata, psoriasis inversa and pustulosis) under therapy with anti-TNF and refractory to at least 12 weeks of topical therapy.
* Written informed consent must be obtained and documented.

Exclusion Criteria:

* IBD patients not treated with anti-TNF therapy
* IBD patients with skin lesions under anti-TNF not refractory to topical therapy
* Patients who previously received anti-interleukin 12/23 (IL12/23) or anti-interleukin 23 therapy
* Patients with history of psoriasis prior to initiation of anti-TNF therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Transcriptomic features | 3 years
  Transcriptomic profile will be established by analysis of the expression of the mRNAs by using Next Generation Sequencing.

SECONDARY OUTCOMES:
Proteomic features | 3 years
  Proteomic profile will be established by using a proximity extension assay from OLINK
Mechanistic changes in psoriasiform skin lesions | 3 years
  Physiological changes that occur with respect to cell types and cytokines will be investigated using immunohistochemistry and cell sorting

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) sharing

REFERENCES:
- [Result] Cleynen I, Van Moerkercke W, Billiet T, Vandecandelaere P, Vande Casteele N, Breynaert C, Ballet V, Ferrante M, Noman M, Assche GV, Rutgeerts P, van den Oord JJ, Gils A, Segaert S, Vermeire S. Characteristics of Skin Lesions Associated With Anti-Tumor Necrosis Factor Therapy in Patients With Inflammatory Bowel Disease: A Cohort Study. Ann Intern Med. 2016 Jan 5;164(1):10-22. doi: 10.7326/M15-0729. Epub 2015 Dec 8. PMID 26641955
- [Result] Cleynen I, Vermeire S. Paradoxical inflammation induced by anti-TNF agents in patients with IBD. Nat Rev Gastroenterol Hepatol. 2012 Sep;9(9):496-503. doi: 10.1038/nrgastro.2012.125. Epub 2012 Jul 3. PMID 22751454
- [Result] Tillack C, Ehmann LM, Friedrich M, Laubender RP, Papay P, Vogelsang H, Stallhofer J, Beigel F, Bedynek A, Wetzke M, Maier H, Koburger M, Wagner J, Glas J, Diegelmann J, Koglin S, Dombrowski Y, Schauber J, Wollenberg A, Brand S. Anti-TNF antibody-induced psoriasiform skin lesions in patients with inflammatory bowel disease are characterised by interferon-gamma-expressing Th1 cells and IL-17A/IL-22-expressing Th17 cells and respond to anti-IL-12/IL-23 antibody treatment. Gut. 2014 Apr;63(4):567-77. doi: 10.1136/gutjnl-2012-302853. Epub 2013 Mar 6. PMID 23468464
- [Result] Grine L, Dejager L, Libert C, Vandenbroucke RE. An inflammatory triangle in psoriasis: TNF, type I IFNs and IL-17. Cytokine Growth Factor Rev. 2015 Feb;26(1):25-33. doi: 10.1016/j.cytogfr.2014.10.009. Epub 2014 Oct 31. PMID 25434285
- [Result] Conrad C, Di Domizio J, Mylonas A, Belkhodja C, Demaria O, Navarini AA, Lapointe AK, French LE, Vernez M, Gilliet M. TNF blockade induces a dysregulated type I interferon response without autoimmunity in paradoxical psoriasis. Nat Commun. 2018 Jan 2;9(1):25. doi: 10.1038/s41467-017-02466-4. PMID 29295985